CLINICAL TRIAL: NCT00979394
Title: Diabetes Care Austria 2009
Brief Title: Evaluation of Diabetes Care at Austrian GPs
Acronym: DCA09
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CAT-DUM-2009/1
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Care at GPs in Austria; Characteristic of diabetes patients at GPs in Austria
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes

SUMMARY:
This registery should show the medical care of patient with Type 2 Diabetes (T2D) at GP-offices. Furthermore data of co morbidities and risk factors should be evaluated. Objectives of this NIS (cross-sectional study) are:

* To evaluate which characteristics or co-morbidities are being existent for patient with T2D at GP level,
* To evaluate representative profile of patient with T2D in Austria,
* To evaluate which medical therapies are used.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type II

Exclusion Criteria:

* Diabetes mellitus type I
* Gestation diabetes
* Induced diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GPs
Sampling Method: Probability Sample
Enrollment: 1513 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Evaluate characteristics or co morbidities being existent for patient with T2D at GP | Once per patient

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Ludvig, Study Chair — General Hospital Vienna; Guntram Schernthaner, Study Chair — Krankenanstalt Rudolfsstiftung